CLINICAL TRIAL: NCT00552578
Title: A Randomized Controlled Trial Testing Buprenorphine as a Treatment in Opiate Dependent Pain Patients
Brief Title: Buprenorphine as a Treatment in Opiate Dependent Pain Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: "Tapering doses" protocol arm was not effective for treatment retention outcome.
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Richard D. Blondell, SUNYBuffalo, Dept Family Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMD0400907A
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Results first posted 2009-07-07 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Opiate Addiction; Refractory Pain
Keywords: drug dependence; substance abuse; substance use disorders; myofascial pain syndrome; neuralgia; back pain
MeSH Terms: conditions — Opioid-Related Disorders; Pain, Intractable; Substance-Related Disorders; Myofascial Pain Syndromes; Neuralgia; Back Pain | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tapering doses of buprenorphine (Active Comparator): Participants assigned to this arm will receive tapering doses of buprenorphine for detoxification.
  Interventions: Drug: buprenorphine/naloxone
- Steady doses of buprenrophine (Experimental): Participants assigned to this arm will receive a steady dose of buprenorphine for maintenance.
  Interventions: Drug: buprenorphine/naloxone

INTERVENTIONS:
Drug: buprenorphine/naloxone — sublingual tablets, 2/0.5 mg, three times a day for one month, twice a day for one month, once a day for one month, then every other day for one month. (dose may be adjusted based on an individual's response)
  Other Names: Suboxone
  Arms: Tapering doses of buprenorphine
Drug: buprenorphine/naloxone — sublingual tablets, 2/0.5 mg, one tablet three times a day for six months (doses may be adjusted based on an individual's response
  Other Names: Suboxone
  Arms: Steady doses of buprenrophine

SUMMARY:
This study is designed to determine if different doses of buprenorphine (either tapering doses or steady doses) are effective in managing chronic, non-cancer pain in individuals who also are addicted to opiate pain medicines.

DETAILED DESCRIPTION:
Context: Some individuals have two conditions: 1) a well-documented pain disorder and 2) clear evidence of a substance use disorder with opiate dependency. It is not known how to manage these patients. In addition to other modalities for the treatment of chronic pain, combination tablets of buprenorphine/naloxone (Suboxone) may be helpful.

Objective: The objective of this study is to determine if the addition of pharmacotherapy with Suboxone to usual care would improve clinical outcome relative to usual care alone.

Design: Randomized control trial.

Setting: The study will be conducted in the out-patient clinics of a tertiary-care teaching hospital.

Participants: The participants will be those who have: 1) a well-documented pain disorder and 2) clear evidence of a substance use disorder with opiate dependency.

Baseline data collected: Data collected at baseline will include (with examples): demographics (age, gender, race), substance use history (type of substances used, duration of use, routes of abuse), type of pain disorder (previous traumatic injury, musculoskeletal, neuropathic), co-existing medical problems (seizures, hepatitis C), prior injuries (accidents, interpersonal violence), prior mental health problems (prior treatment, diagnoses), prior substance abuse treatment (outpatient, inpatient), socioeconomic variables (educational level, occupation, employment history), criminal history (number of arrests and convictions, total amount of time spent in jail or prison), family history (first degree relatives with substance use disorders) and scores on psychometric testing (ASI).

Outcome data: Three main outcome variables will be examined relapse to substance use (as documented by toxicology), quality of life, and successful participation in the pain management program for six months, which included the completion of the study buprenorphine treatment protocols.

Data analyses: Outcome variables will be compared between the two groups using t-tests or chi-square tests as appropriate. A Kaplan-Myer survival analysis will be used to describe participant participation. Predictors of poor outcomes will be identified using a case-control design in which those with poor outcomes (the "cases") will be compared to those with successful outcomes (the "controls") using multivariate techniques (logistic regression).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic refractory pain
* Clinical diagnosis of opiate dependency

Exclusion Criteria:

* unable to pay for medication
* enrolled in a methadone maintenance program
* homelessness
* major mental illness
* pregnant women
* prisoners
* terminal cancer pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Blondell, MD, Principal Investigator — University at Buffalo
Locations (1):
- Erie County Medical Center, Buffalo, New York, United States

REFERENCES:
- [Result] Blondell RD, Ashrafioun L, Dambra CM, Foschio EM, Zielinski AL, Salcedo DM. A Clinical Trial Comparing Tapering Doses of Buprenorphine with Steady Doses for Chronic Pain and Co-existent Opioid Addiction. J Addict Med. 2010 Sep;4(3):140-6. doi: 10.1097/ADM.0b013e3181ba895d. PMID 20959867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 participants recruited Dec 2007 to Apr 2008
Groups:
- Steady Dose of Buprenorphine: Participants assigned to this arm will receive a steady dose of buprenorphine for maintenance.
Period: Overall Study
Arm/Group | Tapering Doses of Buprenorphine | Steady Dose of Buprenorphine
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapering Doses of Buprenorphine | Steady Dose of Buprenorphine | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (6) | 46 (15) | 45 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Relapse to Substance Abuse
Description: Relapse to substance abuse (yes/no) was determined by participant self-report or by a positive urine toxicology.
Time Frame: Six months
Measure: Number; unit: participants
Arm/Group | Tapering Doses of Buprenorphine | Steady Dose of Buprenorphine
Number analyzed (Participants) | 5 | 5
participants | 2 | 4
Statistical Analysis 1: Comparison: Tapering Doses of Buprenorphine vs Steady Dose of Buprenorphine; Intent to treat; Test type: Superiority or Other; p = 0.523, Fisher Exact; Odds Ratio (OR) = 0.17, 95% CI [0.0098 to 2.8215]

2. Secondary Outcome: Number of Participants With Better Overall Quality of Life at Six Months as Compared to Baseline.
Description: Qualitative measure (better/no change/worse) of participant's perception of overall quality of life related to assigned study protocol arm.
Time Frame: Baseline and six months
Population: Reported value (number) was the number who reported a "better" overall quality-of-life to the question: "How would you describe your overall level of function now as compared to the time right before you started the study?" Responses were recorded as: "better," "no change," or "worse."
Measure: Number; unit: Participants
Arm/Group | Tapering Doses of Buprenorphine | Steady Dose of Buprenorphine
Number analyzed (Participants) | 5 | 5
Participants | 4 | 4

3. Secondary Outcome: Treatment Retention.
Description: "Treatment retention" was defined as the completion of the buprenorphine dosing protocol (i.e., tapering doses vs. steady doses).
Time Frame: Six months
Population: Analysis was intent-to-treat.
Measure: Number; unit: Participants
Arm/Group | Tapering Doses of Buprenorphine | Steady Dose of Buprenorphine
Number analyzed (Participants) | 6 | 6
Participants | 0 | 5
Statistical Analysis 1: Comparison: Tapering Doses of Buprenorphine vs Steady Dose of Buprenorphine; Fisher exact test was used and tested the hypothesis that neither group would be more likely to complete the study protocol; Test type: Superiority or Other; p = 0.015, Fisher Exact — No adjustment

ADVERSE EVENTS:
Arm/Group | Tapering Doses of Buprenorphine | Steady Dose of Buprenorphine
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No